CLINICAL TRIAL: NCT02856230
Title: An Efficacy and Safety Study to Evaluate Ranger Drug-eluting Balloon for Below the Knee Angioplasty in Patients With Critical Limb Ischemia
Brief Title: An Efficacy and Safety Study to Evaluate Ranger DEB for BTK Angioplasty in Patients With CLI (RANGER-BTK)
Acronym: RANGER-BTK
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P151101; IDRCB 2016-A00035-46 (Other: Agence Nationale de Securite du Medicament et des Produits de Sante)
Record Dates: First submitted 2016-07-19; First posted 2016-08-04 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Lower Limb Ischemia; Peripheral Vascular Diseases
Keywords: Critical limb ischemia; bellow-the-knee angioplasty; drug-eluting balloon
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranger SL DEB angioplasty (Experimental): patients filling general and angiographic inclusion/exclusion criteria will have an BTK angioplasty using one or several Ranger SL drug-eluting balloons
  Interventions: Device: Ranger SL DEB

INTERVENTIONS:
Device: Ranger SL DEB — BTK angioplasty using Ranger SL DEB
  Other Names: Ranger SL paclitaxel-eluting balloon

SUMMARY:
Endovascular treatment of below the knee disease is a well-established therapy to improve outcomes in patients with critical limb ischemia. Several large cohort studies demonstrated the safety and the efficacy of percutaneous recanalization and angioplasty for distal vessel disease. A successful recanalization of foot artery was related to a higher ulcer healing and a reduction of major amputation. Moreover absence of revascularization in a patient with critical limb ischemia is an independent risk factor for mortality. Despite the introduction of new devices dedicated to below the knee vessel disease treatment, with the development of guides and conical balloons, long term patency outcomes are still poor. Restenosis was observed in more than two thirds of patients within 3 months after angioplasty of tibial arteries with a high target lesions revascularization. These re-interventions are characterized by a higher morbidity and mortality due to several comorbidities associated to these patients. These data confirm the need to obtain more lasting results in order to improve long-term outcomes of these patients.

Recently, the use of drug-eluting balloons (DEB) has revealed an increase in patency after angioplasty of the femoral artery. On the contrary, results for BTK arteries angioplasty have shown controversial results.

The purpose of this study is to evaluate the safety and the efficacy of the Ranger™ SL paclitaxel coated balloon a model of drug eluting balloon in patients with critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria :

* Age ≥18 years and ≤85 years
* Patient signed an approved consent form
* Patient has documented chronic Critical Limb Ischemia (CLI) in the target limb prior to the study procedure with Rutherford Category 4, 5 or 6
* Menopausal or under contraception for women
* Negative serum β-HCG for women of childbearing age

Angiographic Inclusion Criteria :

* Single or multiple lesions with ≥70% diameter stenosis (DS) of different lengths in one or more main below the knee vessels
* Intraluminal recanalization of the target lesion with successful traversal of the target lesion and placement of the guidewire into the distal true lumen
* Reference vessel reference diameter comprised between 2 and 4 mm

Exclusion Criteria:

General non-inclusion criteria:

* Patient with known hypersensitivity to paclitaxel
* Patient unwilling or unlikely to comply with Follow-Up schedule
* Life expectancy <1 year (investigator's appreciation)
* Planned major index limb amputation
* Pregnant or breast feeding women

Angiographic exclusion criteria:

* Significant (≥50% DS) inflow lesion or occlusion in the ipsilateral iliac, superficial femoral or popliteal artery that cannot be treated successfully in the same session
* Previously implanted stent in the target lesions(s)
* Aneurysm in the target vessel
* Acute thrombus in the target limb
* Failure to cross the target lesion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of deaths and major amputations | 6 months
  Number of deaths and major amputations (any amputation above the knee) at 6 months after procedure
Efficacy: Primary patency (no stenosis >50%) of the Target Lesion measured by Quantitative Vascular Angiography (QVA) | 6 months
  Primary patency (no stenosis >50%) of the Target Lesion measured by Quantitative Vascular Angiography (QVA)

SECONDARY OUTCOMES:
Composite of all death and major amputation | 12 months
  Number of deaths and major amputations (any amputation above the knee) at 12 months after procedure
Number of SAEs | 12 months
  Procedure related or contributed total number of SAEs
Number of AEs | 12 months
  Procedure related or contributed total number of AEs
Late Lumen Loss (LLL) | 6 months
  Late Lumen Loss (LLL) of the Target Lesion measured by Quantitative Vascular Angiography (QVA)
Clinically driven Target Lesion Revascularization (TLR) | 6 and 12 months
  Clinically driven TLR is defined as any TLR of the target lesion associated with Deterioration of Rutherford Class and/or increase in size of pre-existing wounds and / or occurrence of a new wound(s)
Amputation Free Survival | 6 and 12 months
Rate of Wound Healing | 6 and 12 months
Quality of Life | 6 and 12 months
  Quality of Life assessed by EQ5D questionnaires
Ulcer diameter | 1, 6 and 12 months
  Ulcer diameter in the target limb
ABI (Ankle-Brachial Index) | 1, 6 and 12 months
  ABI in the target limb
Toe pressure | 1, 6 and 12 months
  Toe pressure in the target limb
Device success rates | Through angioplasty completion
  Percentage of exact deployment of the device according to the instructions for use as documented with suitable imaging modalities
Technical success rates | Through angioplasty completion
  Percentage of successful vascular access, completion of the endovascular procedure and immediate morphological success with less or equal to 50% residual diameter reduction of the treated lesion on completion angiography

CONTACTS AND LOCATIONS:
Overall Officials: Marc SAPOVAL, MD, PhD, Principal Investigator — AP - HP, Hopital Europeen Georges-Pompidou, Paris, France
Locations (1):
- AP-HP - Hopital Europeen Georges-Pompidou Paris, France, Paris, Île-de-France Region, France